CLINICAL TRIAL: NCT00565357
Title: Silicone Earplugs for VLBW Newborns in Intensive Care: Feasibility, Sound Attenuation, and Outcomes From a Randomized Clinical Trial
Brief Title: Silicone Earplugs for VLBW Newborns in Intensive Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R01HD042639-01A3 (NIH)
Record Dates: First submitted 2007-11-27; First posted 2007-11-29 (Estimated); Last update posted 2007-11-29 (Estimated); Status verified 2007-11

CONDITIONS: Postnatal Growth
Keywords: Postnatal Growth; Postnatal Development; Noise; Neonatal Intensive Care Unit

ARMS (2):
- E (Experimental)
  Interventions: Device: Silicone Earplugs
- C (No Intervention)
  Interventions: Other: Control

INTERVENTIONS:
Device: Silicone Earplugs — Silicone earplugs worn from within 1 week of birth through 35 weeks post-menstrual age or hospital discharge, whichever came first
  Arms: E
Other: Control — Standard care in the neonatal intensive care unit
  Arms: C

SUMMARY:
The purpose of this study was to determine the effects of individual noise reduction using silicone earplugs for very low birthweight newborns in neonatal intensive care on growth and development. The study hypothesis was that newborns who were randomized to the earplug group would be heavier than controls at 34 weeks post-menstrual age.

ELIGIBILITY:
Inclusion Criteria:

* birthweight between 401 and 1500 grams
* less than 1 week of age
* parental informed consent
* availability of research personnel

Exclusion Criteria:

* terminal illness
* congenital anomalies
* syndromes associated with hearing loss

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2002-06; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Weight | 34 weeks post-menstrual age

SECONDARY OUTCOMES:
Length of stay in neonatal intensive care | hospital discharge
Time on mechanical ventilator | hospital discharge
Weight | 18 - 22 months of age
Length | 18 - 22 months of age
Frontal-occipital circumference | 18 - 22 months of age
Bayley Mental Developmental Index | 18 - 22 months of age
Bayley Psychomotor Developmental Index | 18 - 22 months of age
ABR Hearing Screen | hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Robert E Lasky, PhD, Principal Investigator — University of Texas Medical School at Houston

REFERENCES:
- [Derived] Abou Turk C, Williams AL, Lasky RE. A randomized clinical trial evaluating silicone earplugs for very low birth weight newborns in intensive care. J Perinatol. 2009 May;29(5):358-63. doi: 10.1038/jp.2008.236. Epub 2009 Feb 5. PMID 19194455